CLINICAL TRIAL: NCT00267306
Title: A Phase 1/2, Partially Randomized, Open-Label Study of Visilizumab in Patients With Severe Ulcerative Colitis Refractory to Intravenous Corticosteroids
Brief Title: Ulcerative Colitis Study: Study of Visilizumab in Patients With Severe Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 291-408
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Severe Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of visilizumab in patients with severe ulcerative colitis that has failed to respond to steroid therapy.

What is visilizumab?

Visilizumab is an antibody designed to reduce inflammation. Antibodies are proteins that are normally made by the immune system to help defend the body from infections and other foreign substances. Visilizumab is thought to selectively affect the immune system to decrease inflammation and, in doing so, it may prevent damage to the intestine caused by ulcerative colitis.

Who can participate in this study?

The target population for this study is adults with severe ulcerative colitis that has resisted intravenous (IV) steroids. This study is open to patients with the following characteristics:

* 16-70 year olds
* A diagnosis of ulcerative colitis verified by colonoscopy or barium enema performed within 36 months prior to study entry
* Active disease despite ongoing treatment with steroids

How is this study conducted?

Eligible participants will be administered visilizumab as one daily injection on two consecutive days. All medication and study-related care, except for the costs of in-patient hospitalization, are provided to qualified participants at no cost. This includes all visits, examinations and laboratory work.

How does one get more information?

This study is currently enrolling patients at hospitals and clinics in North America and Europe. For more information on the study or how to participate in it, please call 1-800-772-0482, email InfoCenter@pdl.com or visit www.IBDtrials.com.

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* 16 -70 year olds
* A diagnosis of ulcerative colitis verified by colonoscopy or barium enema performed within 36 months prior to study entry
* Active disease despite ongoing treatment with IV steroids

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of visilizumab in patients with severe ulcerative colitis that is resistant to intravenous steroids

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Inflammatory Bowel Disease Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Medical College of Cornell, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - UPHS/Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

REFERENCES:
- [Derived] Baumgart DC, Targan SR, Dignass AU, Mayer L, van Assche G, Hommes DW, Hanauer SB, Mahadevan U, Reinisch W, Plevy SE, Salzberg BA, Buchman AL, Mechkov GM, Krastev ZA, Lowder JN, Frankel MB, Sandborn WJ. Prospective randomized open-label multicenter phase I/II dose escalation trial of visilizumab (HuM291) in severe steroid-refractory ulcerative colitis. Inflamm Bowel Dis. 2010 Apr;16(4):620-9. doi: 10.1002/ibd.21084. PMID 19714757